CLINICAL TRIAL: NCT01300572
Title: A Study Evaluating Escalating Doses of 90Y-DOTA-BC8 (Anti-CD45) Antibody Followed by Allogeneic Stem Cell Transplantation for High-Risk Acute Myeloid Leukemia (AML) Acute Lymphoblastic Leukemia (ALL), or Myelodysplastic Syndrome (MDS)
Brief Title: Yttrium-90 Anti-CD45 Monoclonal Antibody BC8 Followed by Donor Stem Cell Transplant in Treating Patients With High-Risk AML, ALL, or MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2468.00; NCI-2011-00150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2468.00A; 2468; 2468.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2011-02-15; First posted 2011-02-21 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Chronic Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Indium; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Y-90-BC8 & Allogeneic Transplant (Experimental): PREPARATIVE REGIMEN: Patients receive 90Y-BC8 via central line on approximately day -12, fludarabine phosphate IV over 30 minutes on days -4 to -2, and 2 Gy TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive mycophenolate mofetil PO or IV every 12 hours on days 0-27 (for patients with related donors) or every 8 hours on days 0-40 with taper to day 96 (for patients with unrelated donors). Patients also receive cyclosporine PO or IV every 12 hours on days -3 to 56 (for patients with related donors) or 100 (for patients with unrelated donors) with taper to day 180.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Biological: Indium In 111 Anti-CD45 Monoclonal Antibody BC8; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Total-Body Irradiation; Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSC or bone marrow transplant
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Indium In 111 Anti-CD45 Monoclonal Antibody BC8 — Given IV (dosimetric dose)
  Other Names: In 111 MOAB BC8; In 111 Monoclonal Antibody BC8; Indium In 111 Monoclonal Antibody BC8; monoclonal antibody BC8, indium In 111
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation
Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8 — Given via central line (therapeutic dose)
  Other Names: 90Y Anti-CD45 MoAb BC8

SUMMARY:
This phase I trial studies the side effects and maximum tolerated dose of yttrium Y 90 anti-cluster of differentiation 45 (CD45) monoclonal antibody BC8 (90Y-BC8) followed by donor stem cell transplant in treating patients with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or myelodysplastic syndrome (MDS) that is likely to come back or spread. Giving chemotherapy drugs, such as fludarabine phosphate (FLU), and total-body irradiation (TBI) before a donor peripheral blood stem cell (PBSC) or bone marrow transplant helps stop the growth of cancer or abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. Radiolabeled monoclonal antibodies, such as 90Y-BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving FLU, 90Y-BC8, and TBI before the transplant together with cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of radiation delivered via 90Y-DOTA-BC8 (90Y-BC8) when combined with FLU and 2 Gy TBI as a preparative regimen for patients aged >= 18 with advanced AML, ALL, and high-risk MDS.

SECONDARY OBJECTIVES:

I. To determine disease response and duration of remission.

II. To determine the rates of engraftment and donor chimerism resulting from this combined preparative regimen, and to correlate level of donor chimerism with estimated radiation doses delivered to hematopoietic tissues via antibody.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive 90Y-BC8 via central line on approximately day -12 and FLU intravenously (IV) over 30 minutes on days -4 to -2.

TRANSPLANTATION: Patients undergo TBI followed by allogeneic PBSC or bone marrow transplant on day 0.

GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive mycophenolate mofetil orally (PO) or IV every 12 hours on days 0-27 (for patients with related donors) or every 8 hours on days 0-40 with taper to day 96 (for patients with unrelated donors). Patients also receive cyclosporine PO or IV every 12 hours on days -3 to 56 (for patients with related donors) or 100 (for patients with unrelated donors) with taper to day 180.

After completion of study treatment, patients are followed up at 6, 9, 12, 18, and 24 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced AML, ALL or high-risk MDS meeting one of the following descriptions:

  * AML or ALL beyond first remission (i.e., having relapsed at least one time after achieving remission in response to a treatment regimen)
  * AML or ALL representing primary refractory disease (i.e., having failed to achieve remission at any time following one or more prior treatment regimens)
  * AML evolved from myelodysplastic or myeloproliferative syndromes; or
  * MDS expressed as refractory anemia with excess blasts (RAEB) or chronic myelomonocytic leukemia (CMML) by French-American-British (FAB) criteria
* Patients not in remission must have CD45-expressing leukemic blasts; patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to non-malignant cells which make up >= 95% of nucleated cells in the marrow)
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must have an estimated creatinine clearance greater than 50/ml per minute (serum creatinine value must be within 28 days prior to registration)
* Bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine transaminase (ALT) < 2 times the upper limit of normal
* Eastern Cooperative Oncology Group (ECOG) =< 2 or Karnofsky >= 70
* Patients must have an expected survival of > 60 days and must be free of active infection
* Patients must have an human leukocyte antigen (HLA)-identical sibling donor or an HLA-matched unrelated donor who meets standard Seattle Cancer Care Alliance (SCCA) and/or National Marrow Donor Program (NMDP) or other donor center criteria for PBSC or bone marrow donation, as follows:

  * Related donor: related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1; phenotypic identity must be confirmed by high-resolution typing
  * Unrelated donor:

    * Matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; OR mismatched for a single allele without antigen mismatching at HLA-A, B or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * Doors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before hematopoietic cell transplant (HCT); if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with and HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
    * Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch; i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Donors must meet HLA matching criteria and standard SCCA and/or National Marrow Donor Program (NMDP) or other donor center criteria for PBSC or bone marrow donation

Exclusion Criteria:

* Circulating human anti-mouse antibody (HAMA)
* Prior radiation to maximally tolerated levels to any critical normal organ, or > 20 Gy prior radiation to large areas of the bone marrow (e.g., external radiation therapy to whole pelvis)
* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Left ventricular ejection fraction < 35%
* Corrected diffusion lung capacity of carbon monoxide (DLCO) < 35% or receiving supplemental continuous oxygen
* Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Patients who are known to be seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures
* Active central nervous system (CNS) leukemia at time of treatment
* Women of childbearing potential who are pregnant (beta-human chorionic gonadotropin positive [HCG+]) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Inability to understand or give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Vo P, Gooley TA, Rajendran JG, Fisher DR, Orozco JJ, Green DJ, Gopal AK, Haaf R, Nartea M, Storb R, Appelbaum FR, Press OW, Pagel JM, Sandmaier BM. Yttrium-90-labeled anti-CD45 antibody followed by a reduced-intensity hematopoietic cell transplantation for patients with relapsed/refractory leukemia or myelodysplasia. Haematologica. 2020 Jun;105(6):1731-1737. doi: 10.3324/haematol.2019.229492. Epub 2019 Oct 3. PMID 31582553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol is open to participants age 18 and above, of either gender and any race/ethnicity. The study is looking at the use of Y-90-DOTA-BC8 in conjunction with a standard reduced-intensity transplant regimen.
Groups:
- Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant): PREPARATIVE REGIMEN: Patients receive 90Y-BC8 via central line on approximately day -12, fludarabine phosphate IV over 30 minutes on days -4 to -2, and 2 Gy TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive mycophenolate mofetil PO or IV every 12 hours on days 0-27 (for patients with related donors) or every 8 hours on days 0-40 with taper to day 96 (for patients with unrelated donors). Patients also receive cyclosporine PO or IV every 12 hours on days -3 to 56 (for patients with related donors) or 100 (for patients with unrelated donors) with taper to day 180.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic bone marrow transplant
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or bone marrow transplant
  Cyclosporine: Given PO or IV
  Fludarabine Phosphate: Given IV
  Indium In 111 Anti-CD45 Monoclonal Antibody BC8: Given IV (dosimetric dose)
Period: Overall Study
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Started | 16
Completed | 15
Not Completed | 1
Not completed — HAMA + post dosimetry | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant): Study participants will receive an infusion of 0.5 mg/kg of ideal body weight of DOTA-BC8 trace labeled with ~5-10 mCi of Indium-111 to evaluate biodistribution and calculate the radiation absorbed doses to major organs and the whole body. The subsequent therapy infusion of Yttrium-90-DOTA-BC8 will deliver an amount of Yttrium-90 calculated not to exceed the target dose to the critical normal organ receiving the highest radiation dose. The therapy dose will be administered on approximately day -12 of the preparative regimen, which will typically be approximately 1 to 2 weeks after the biodistribution dose.
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The MTD of Radiation Delivered Via 90Y-DOTA-BC8 When Combined With FLU and 2 Gy TBI as a Preparative Regimen for Patients Aged ≥ 18 With Advanced AML, ALL, and High-risk MDS.
Description: The MTD will be defined as the dose that is associated with a true DLT rate of 25%. The highest dose achieved was 28 Gy but none of the patients experienced a DLT. Thus, the MTD was not reached.
Time Frame: Within the first 30 days following transplant
Population: Study participants who completed the study regimen.
Measure: Number; unit: Gy
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
Gy | 28

2. Secondary Outcome: Achievement of Remission
Description: Number of participants who are in complete remission (CR) 4 weeks after transplant. CR is defined as complete resolution of all signs of myelodysplasia or leukemia for at least 4 weeks with all of the following:
  1. Normal bone marrow with blasts <5% with normal cellularity, normal megakaryopoiesis, > 15% erythropoiesis and > 25% granulocytopoiesis
  2. Normalization of blood counts (no blasts, platelets > 100000/mm3, granulocytes >1500/mm3)
  3. No extramedullary disease.
Time Frame: 4 weeks after transplant
Population: Study participants who completed the study regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
Participants | 13

3. Secondary Outcome: Disease-free Survival
Description: Number of study participants who are alive and remains in complete remission after transplant.
Time Frame: 100 days after transplant
Population: Study participants who completed study regimen and in CR after transplant.
Measure: Number; unit: participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
participants | 7

4. Secondary Outcome: Duration of Remission
Description: Median time to relapse after achieving complete remission (CR). CR is defined as complete resolution of all signs of myelodysplasia or leukemia for at least 4 weeks with all of the following:
  1. Normal bone marrow with blasts <5% with normal cellularity, normal megakaryopoiesis, > 15% erythropoiesis and > 25% granulocytopoiesis
  2. Normalization of blood counts (no blasts, platelets > 100000/mm3, granulocytes >1500/mm3)
  3. No extramedullary disease.
  Relapse Criteria:
  1. After CR: >5% blasts in the bone marrow and/or peripheral blood
  2. After partial remission (PR): increase of blasts cells in the marrow to >50% of those during PR
  3. Extramedullary disease confirmed cytologically or histologically.
Time Frame: 1 year
Population: Study participants who relapsed after achieving complete remission after transplant.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 13
days | 213 [69 to 351]

5. Secondary Outcome: Estimation of Absorbed Radiation Doses to Normal Organs, Marrow and Tumor
Description: The amount of energy absorbed per unit weight of the organ or tissue is called absorbed dose and is expressed in units of gray (Gy). One gray dose is equivalent to one joule radiation energy absorbed per kilogram of organ or tissue weight.
Time Frame: Approximately day -20 to day -12 prior to transplant
Population: All study participants who completed the study regimen.
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
Gy
  Average absorbed dose to the marrow | 11.4 (9.2)
  Average absorbed dose to the liver | 17.2 (6.8)
  Average abosorbed dose total body | 3.1 (5.7)
  Average absorbed dose to the spleen | 70 (43)

6. Secondary Outcome: Overall Survival
Description: Number of participants who are still alive after transplant with or without disease.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
Participants | 7

7. Secondary Outcome: Rates of Acute GvHD
Description: Number of participants who developed acute GVHD post-transplant, aGVHD stages:
  Skin: a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Up to 84 days post-transplant
Population: Overall number of participants analyzed is 14 because one patient died prior to d+84 after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 14
Participants
  Grade 0 acute GVHD | 4
  Grade I acute GVHD | 1
  Grade II acute GVHD | 6
  Grade III acute GVHD | 2
  Grade IV acute GVHD | 1

8. Secondary Outcome: Rates of Donor Chimerism
Description: Number of participants who has 100% donor chimerism within 100 days after transplant
Time Frame: Up to 100 days post-transplant
Population: Overall number of participants analyzed is 14 because one patient died prior to d+84 after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 14
Participants | 14

9. Secondary Outcome: Rates of Engraftment
Description: Average number of days to ANC >= 500 after transplant
Time Frame: Up to 84 days post-transplant
Population: Study participants with an ANC <= to 500 after transplant
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 14
days | 16 (6.0)

10. Secondary Outcome: Rates of Non-relapse Mortality
Description: Transplant-related deaths within 100 days after transplant
Time Frame: Within the first 100 days following transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
Number analyzed (Participants) | 15
Participants
  Severe refractory GVHD | 1
  Bacterial infection | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) will be monitored and recorded in study-specific case report forms (CRFs) from the time of first exposure to an investigational agent (i.e., the start of the Indium-111-DOTA-BC8 infusion) through day +100 after transplant or through discharge prior to that date from the SCCA system to the care of the patient's primary physician.
Description: Non-hematologic adverse events of ≥ grade 3, possibly related events of grade 2 that have not previously been observed with components of the study regimen, and all serious adverse events will be captured in protocol-specific case report forms. Beyond day +100, disease progression, development of secondary malignancies, and survival only will be collected.
Groups:
- Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant): PREPARATIVE REGIMEN: Patients receive 90Y-BC8 via central line on approximately day -12, fludarabine phosphate IV over 30 minutes on days -4 to -2, and 2 Gy TBI on day 0. TRANSPLANTATION: Patients undergo allogeneic PBSC or bone marrow transplant on day 0.
Arm/Group | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant)
All-Cause Mortality (participants affected / at risk) | 5/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant) (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Vomiting (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Skin infection (Infections and infestations) | 1 — Cellulitis
Hypokalemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (90Y-BC8, Allogeneic PBSC or Bone Marrow Transplant) (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis, oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 1
Edema limbs (General disorders) | 4
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 6
Fever (General disorders) | 2
Allergic reaction (Immune system disorders) | 6
Coag negative staph infection (Infections and infestations) | 1
CMV reactivation (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection - Rhinovirus (Infections and infestations) | 1
Upper respiratory infection - Rhinorrea (Infections and infestations) | 1
Upper respiratory infection - Metapneumovirus (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, trunk (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The highest dose achieved was 28 Gy but none of the patients experienced a DLT. Thus, the MTD was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT01300572/Prot_SAP_000.pdf